CLINICAL TRIAL: NCT04987437
Title: Prospective Observational Case Series Analysing Outcomes of Primary Hip Arthroplasty With a Short Cemented Stem (Friendly Short)
Brief Title: Prospective Observational Case Series of Primary Hip Arthroplasty With a Short Cemented Stem (Friendly Short)
Status: Completed | Type: Observational
Sponsor: Limacorporate S.p.a (Industry)
Responsible Party: Sponsor
Other Study IDs: H-02
Record Dates: First submitted 2021-07-27; First posted 2021-08-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Total Hip Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Friendly short stem — Total Hip Arthroplasty with Friendly Short stem

SUMMARY:
Post-marketing observational case series to analyse the functional recover and radiographic outcomes in terms of implant stability and survivorship of primary hip arthroplasty with Friendly short cemented stem.

DETAILED DESCRIPTION:
The aim of this case series is to verify the functional recover and radiographic outcomes of primary hip arthroplasty with Friendly short cemented stem.

This is a post-marketing clinical investigation, the product on study is CE marked and used according to the intended use.

It is a national, mono-centre, prospective, observational case series on 100 patients in 1 site.

Primary endpoint is to investigate clinical progression of patients with THA with Friendly short stem from baseline to 1-year follow-up.

The secondary endpoint is to evaluate implant stability and survivorship of implants up to 5 years Follow-up.

The evaluation has an internal control because the assessment of post-treatment data is compared to baseline measurements (pre-operative clinical analysis and radiographic analysis at discharge).

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders;
* Patients of all ages, but > 18 years old;
* Patients with primary and secondary coxarthrosis;
* Patients with rheumatoid arthritis;
* Patients with avascular necrosis;
* Patients with neck (not diaphyseal) fractures;
* Patients requiring a primary hip arthroplasty.

Exclusion Criteria:

* Patients requiring a revision of a previous stem;
* Patients with proven active or suspicious infections;
* Patients with known hypersensitivity to used materials;
* Patients with known active neoplastic or metastatic diseases;
* Patients with significant neurological or musculoskeletal disorders that may affect functional recover;
* Patients with proven haemophilic disease;
* Patients with unwilling or unable to comply with rehabilitation or inability to return for follow-up visits;
* Women with pregnancy or childbearing capacity or breast-feeding;
* Subjects already enrolled in other clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring a primary hip arthroplasty, due to primary and secondary coxarthrosis, avascular necrosis, rheumatoid arthritis, neck (but not diaphyseal) fractures
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-05-02 (Actual); Primary Completion 2013-12-06 (Actual); Study Completion 2018-11-06 (Actual)

PRIMARY OUTCOMES:
change in percentage of the results of the absolute and weighted (age, gender) Harris Hip Score score from baseline to 1 year | up to 5 years FU
Change in percentage of the results of the Oxford Hip Score baseline to 1 year | up to 5 years FU
Change in Range Of Motion from baseline to 1 year. | up to 5 years FU

SECONDARY OUTCOMES:
Radiographic stability | up to 5 years FU
  rate of signs of subsidence > 2mm or tilting
Rate of failure | up to 5 years FU
  rate or revisions, loosening, failure of cement-stem interface, cement cracks, any definite change in the position of components
Any possible adverse event or complication | up to 5 years FU

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Clinico Sant'Anna, Brescia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marega L, Gnagni P, Marega C, Marega F. Mid-term outcomes after primary total hip arthroplasty with a cemented short stem in an elderly patient cohort. Arch Orthop Trauma Surg. 2024 Dec 27;145(1):96. doi: 10.1007/s00402-024-05734-3. PMID 39729135